CLINICAL TRIAL: NCT02148276
Title: Improving Identification of Social Harm Among Substance Abusers in HIV Trials
Status: Completed | Type: Observational
Sponsor: Treatment Research Institute (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Organization: Public Health Management Corporation (Other)
Other Study IDs: 1408; R21DA036407 (NIH)
Record Dates: First submitted 2014-05-23; First posted 2014-05-28 (Estimated); Last update posted 2023-03-28 (Actual); Status verified 2023-03

CONDITIONS: Social Harms in Substance Users in HIV Trials; Audio Computer Assisted Self-administered Questionnaire
Keywords: Social harm detection; Instrument development; HIV-related clinical trials; Substance abuse; Research participation
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Research Participants: All participants will complete two measures of social harm at monthly research appointments for a three month period. The social harms assessments will be (1) the ACASI-SHQ that was developed in Phase 1 and (2) the HIV Vaccine Trials Network (HVTN) Social Impact Assessment.

SUMMARY:
This two-phased project will develop a comprehensive, audio computer assisted self-administered interview social harm questionnaire (ACASI-SHQ) that will allow researchers to more easily identify and monitor social harms experienced by substance abusers participating in HIV-related trials. The ACASI-SHQ will (1) reduce the likelihood of socially desirable responding, (2) include items with high levels of specificity to increase the likelihood of identifying social harms (construct validity), and (3) utilize a self-interview format that will increase the likelihood of its adoption by HIV researchers. The investigators will then evaluate its feasibility, acceptability, and preliminary utility and construct validity in an ongoing HIV-related trial.

DETAILED DESCRIPTION:
Most clinical trials do not regularly monitor for negative social harms experienced by participants in any systematic way. Participation in HIV trials often places participants at a heightened risk of oppression, discrimination, and victimization. These risks may be compounded when participants are substance abusers. Although foreseen risks are generally outlined in the consent form and monitored throughout the study, many social harms are unforeseen and, consequently, are not discussed or monitored. Without systematic monitoring, the majority of social harms likely go undetected. Recognizing the high level of social harm that may arise as a result of participation in HIV vaccine trials, several National Institute of Allergy and Infectious Diseases (NIAID)-sponsored groups began to incorporate general assessments to measure the social impact of research participation in HIV vaccine trials. Although this has provided a preliminary model for monitoring social harms in clinical research, the assessments have several shortcomings that limit their reliability, validity, and utility. In general, they are administered in an interview format that may be cumbersome to the research team. Furthermore, participants may feel uncomfortable or reluctant to report social harms directly to the interviewer, resulting in inaccuracies or underreporting of negative events. Interview items generally address large classes of behavior rather than specific behaviors, reducing the sensitivity and construct validity of the assessments, and questions used across agencies are not standardized. Finally, these assessments do not include harms specific to substance use, a major risk factor for HIV/AIDS transmission. The two-phased project aims to improve the collection of social harms among HIV trial participants by developing a comprehensive, audio computer assisted self-administered interview social harm questionnaire (ACASI-SHQ) that will allow researchers to more easily identify and monitor social harms experienced by substance abusers participating in HIV trials. The proposed study will proceed in two phases. In Phase 1, the investigators will develop the ACASI Social Harm Questionnaire (SHQ). In Phase 2, the investigators will conduct a controlled study to evaluate its acceptability, feasibility, and utility and construct validity.

During Phase 1 the investigators will first conduct a systematic literature review to identify existing tools that researchers currently use to measure social harm or impact experienced by research participants. In addition, the investigators will survey 100 researchers who are currently conducting National Institutes of Health (NIH)-funded HIV-related trials involving substance abusers. The sample will be randomly selected from a pool of researchers meeting this criterion identified through the NIH RePORTER database. The brief telephone survey will include questions about methods used to collect data on social harm including specific questions asked, mode of administration, frequency of assessment, perceived ease of data collection, and concerns related to the assessment. During this phase the investigators will also conduct a focus group with 10 former research participants to gather information about their experiences and perceptions of social harm in HIV-related research trials. The research team in collaboration with a multidisciplinary panel of experts will draft a beta-version of the SHQ content and format. The expert panel will also assist in identifying an optimal trial in which to test the finalized instrument in the second phase of the study. Finally, the investigators will conduct a protocol analysis of the beta-version through interviews with 20 individuals who are currently enrolled in an ongoing National Institute of Drug Abuse (NIDA)-funded HIV prevention trial being conducted by the investigators. This is intended to ensure that items are correctly and similarly understood by subjects, and to provide insight into better methods of phrasing or structuring questions and response options to properly convey their meaning. Upon completion of the protocol analysis, the revised instrument will be finalized by the investigators, programmed into the ACASI format, beta-tested by the research team, and critically reviewed by our expert panel before the final programming of the ACASI-SHQ is completed.

During Phase 2, we will conduct a pilot study to evaluate the acceptability, feasibility, and utility and construct validity of the ACASI-SHQ. Individuals consenting to the host study will be offered the opportunity to participate in the pilot study, and they will receive a manualized written informed consent procedure. We will enroll a total of 80 individuals into the pilot study. All participants will complete two measures of social harm at monthly research appointments for a three month period. The social harms assessments will be (1) the ACASI-SHQ that was developed in Phase 1 and (2) the HIV Vaccine Trials Network (HVTN) Social Impact Assessment. At each appointment, the order in which the instruments are delivered will be counterbalanced to control for carryover effects. At the end of Phase 2, host study research team will complete the ACASI-SHQ Feasibility and Acceptability Questionnaire. Additionally, the PI and Co-I will conduct a focus group with the research team to collect qualitative data on the feasibility, acceptability, and perceived benefits of the ACASI-SHQ and information to guide its future implementation.

The recruitment, study design, conditions, arms, interventions, and eligibility criteria sections of this record reflect the involvement of the 80 participants who will participate in Phase 2 pilot testing of the ACASI-SHQ.

ELIGIBILITY:
Inclusion Criteria:

* Currently participating in an HIV-related trial
* Current or former substance abusers
* 18 years of age or older

Exclusion Criteria:

* Unable to give competent informed consent
* Involvement in the study would negatively affect the participant's health or safety

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We anticipate that the sample will be representative of the populations in our ongoing trials of clients with substance use disorders and of the substance abuse treatment population, which is approximately 70% male, 60% African-American, 35% Caucasian, and 30% Hispanic. This distribution is similar to the gender and racial distributions of publicly funded drug abuse treatment patients in Philadelphia and other large cities located in Mid-Atlantic States.
Sampling Method: Non-Probability Sample
Enrollment: 79 (Actual)
Dates: Start 2015-05; Primary Completion 2017-04-04 (Actual); Study Completion 2017-04-04 (Actual)

PRIMARY OUTCOMES:
Acceptability to participants | 3 months
  Evaluate the acceptability of the ACASI-SHQ to clients using a modified version of the well-validated Client Satisfaction Questionnaire.
Feasibility and acceptability to research staff | 22 Months
  Assess the host study research team's perceptions of the ACASI-SHQ's acceptability and feasibility using the the ACASI-SHQ Feasibility and Acceptability Questionnaire. We will also hold a focus group with the host study research team to collect qualitative data on the feasibility, acceptability, and perceived benefits of the ACASI-SHQ and information to guide its future implementation.

SECONDARY OUTCOMES:
Utility and construct validity | 12 months
  Evaluate the preliminary utility and construct validity of the ACASI-SHQ by comparing the number of social harms it identifies to the number identified using the HVTN social impact assessment. Improved construct validity would be demonstrated if more harms were identified using the ACASI-SHQ than the HVTN social impact assessment.

CONTACTS AND LOCATIONS:
Overall Officials: David S Festinger, Ph.D., Principal Investigator — Treatment Research Institute
Locations (1):
- Treatment Research Institute, Philadelphia, Pennsylvania, United States

REFERENCES:
- See also: Treatment Research Institute — http://www.tresearch.org/